CLINICAL TRIAL: NCT03078608
Title: A Pilot Study of a Mobile/Online-based Mindfulness Intervention for Cancer Patients and Caregivers
Brief Title: POEM (Practice Of Embracing Each Moment) STUDY
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CN-17-2851
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Distress; Cancer; Chemotherapy Effect
Keywords: anxiety; quality of life; mindfulness; meditation; depression
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Experimental): Participants in the intervention arm will receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks.
  Interventions: Behavioral: Mindfulness meditation program (administered via mobile app)
- Active control arm (Active Comparator): Participants in this arm will receive access to a mobile app-based/online progressive muscle relaxation (PMR) program and asked to practice PMR daily for 8 weeks.
  Interventions: Behavioral: Progressive muscle relaxation (via mobile app)
- Wait list control arm (Other): Participants in the wait list control arm will also receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks, but they will not receive access to the program until after the intervention group completes the intervention (8 weeks later).
  Interventions: Behavioral: Mindfulness meditation program (administered via mobile app)

INTERVENTIONS:
Behavioral: Mindfulness meditation program (administered via mobile app) — Mobile app-based/online mindfulness meditation program
  Arms: Intervention arm; Wait list control arm
Behavioral: Progressive muscle relaxation (via mobile app) — Mobile app-based/online progressive muscle relaxation program
  Arms: Active control arm

SUMMARY:
A cancer diagnosis is extremely stressful, emotionally challenging, and often life-altering for both patients and their loved ones. Although more than one-third of patients experience distress, doctors are typically at a loss as to how to help patients and their families manage these emotional challenges. Mindfulness-based programs, including meditation, are offered at major medical centers in the US and have been found to help reduce stress and improve quality of life among cancer patients. However, these classes often require 30+ hours of in-person instruction over 8 weeks, which is neither practical nor feasible for patients undergoing chemotherapy due to side effects and scheduling conflicts.

This study will test whether an 8-week mobile app-based mindfulness program is accepted and useful for patients who have recently received chemotherapy and their loved ones. It will also test whether it is feasible to randomize participants into three groups: intervention, active control (receiving progressive muscle relaxation through the same app) and a wait list control group (will receive the meditation intervention 8 weeks later), so that a future study can test whether mindfulness intervention can help reduce stress and improve quality of life. Because many Americans own smartphone or tablet, an app that can teach stress reduction techniques at home or at infusion clinics has great potential to address emotional needs that providers often cannot.

The study will also include caregivers of patients who have recently received chemotherapy as research has shown that caregivers tend to show high levels of stress and depression and worse physical health compared to non-caregivers. The negative effects of caregiving are most pronounced in caregivers of patients with cancer. However, little support is directed to caregivers as most medical attention goes toward the patients. The patient-caregiver relationship may serve as a source of mutual support and a surrogate for community, which is traditionally considered to be an essential ingredient for sustaining mindfulness practices.

If this study is successful, it will justify a larger trial to determine if use of a mindfulness app is effective in reducing stress and improving quality of life for cancer patients and caregivers. If effective, this low-cost stress reduction strategy could be distributed and used for all types and stages of cancer patients and their caregivers, anywhere, any time, helping to improve the quality of life of the many individuals affected by cancer.

ELIGIBILITY:
Inclusion Criteria:

* active member of Kaiser Permanente Northern California
* a diagnosis of cancer, and currently undergoing chemotherapy or completed chemotherapy in the past 6 months at time of recruitment
* English literacy/fluency, access to a smartphone, a tablet (e.g., iPad) or a computer with internet
* Caregivers: a partner, other family member, or a close friend who identify him/herself as the patient's primary unpaid caregiver. English literacy/fluency, access to a smartphone, a tablet (e.g., iPad) or a computer with internet access

Exclusion Criteria:

* Deafness
* severe mental illness
* Hospital Anxiety and Depression Scale score <8 or >14 on either anxiety or depression scale (patient only)
* current stress reduction practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ai Kubo, PhD, Principal Investigator — Kaiser Permanente Northern California, Division of Research
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kubo A, Kurtovich E, McGinnis M, Aghaee S, Altschuler A, Quesenberry C Jr, Kolevska T, Avins AL. A Randomized Controlled Trial of mHealth Mindfulness Intervention for Cancer Patients and Informal Cancer Caregivers: A Feasibility Study Within an Integrated Health Care Delivery System. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419850634. doi: 10.1177/1534735419850634. PMID 31092044

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm--PATIENTS: Patient-participants in the intervention arm will receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks.
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Wait List Control Arm--PATIENTS: Patient-participants in the wait list control arm will also receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks, but they will not receive access to the program until after the intervention group completes the intervention (8 weeks later).
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Intervention Arm--CAREGIVERS: Caregiver-participants in the intervention arm will receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks.
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Wait List Control Arm--CAREGIVERS: Caregiver-participants in the wait list control arm will also receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks, but they will not receive access to the program until after the intervention group completes the intervention (8 weeks later).
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
Period: Overall Study
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Started | 54 | 43 | 17 | 14
Completed | 40 | 32 | 13 | 13
Not Completed | 14 | 11 | 4 | 1
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 8 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS | Total
Number analyzed (Participants) | 54 | 43 | 17 | 14 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.1) | 56.7 (14.7) | 57.1 (17.4) | 58.2 (18.6) | 58.0 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 9 | 9 | 84
  Male | 21 | 10 | 8 | 5 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 3 | 0 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 0 | 1 | 7
  White | 36 | 27 | 15 | 9 | 87
  More than one race | 8 | 9 | 2 | 2 | 21
  Unknown or Not Reported | 1 | 3 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 36 | 27 | 15 | 9 | 87
  Race: African American | 5 | 1 | 0 | 1 | 7
  Race: Asian | 4 | 3 | 0 | 2 | 9
  Race: Other | 8 | 9 | 2 | 2 | 21
  Race: Unknown/not reported | 1 | 3 | 0 | 0 | 4
Education [Count of Participants; unit: Participants]
  Some college or less | 18 | 19 | 6 | 5 | 48
  College graduate | 15 | 18 | 6 | 4 | 43
  Postgraduate degree | 20 | 6 | 5 | 5 | 36
  Missing | 1 | 0 | 0 | 0 | 1
Income [Count of Participants; unit: Participants]
  Less than $75 000 | 11 | 21 | 2 | 3 | 37
  $75 000 to $99 999 | 7 | 5 | 3 | 3 | 18
  $100 000 to $149 999 | 18 | 8 | 5 | 1 | 32
  $150 000 or more | 12 | 5 | 5 | 3 | 25
  Missing | 6 | 4 | 2 | 4 | 16
Cancer type [Count of Participants; unit: Participants]
  Breast | 13 | 15 | 0 | 0 | 28
  Hematologic | 13 | 8 | 0 | 0 | 21
  Gastrointestinal | 10 | 2 | 0 | 0 | 12
  Genitourinary | 5 | 7 | 0 | 0 | 12
  Head and neck | 4 | 1 | 0 | 0 | 5
  Skin | 3 | 1 | 0 | 0 | 4
  Lung | 0 | 3 | 0 | 0 | 3
  Other | 2 | 1 | 0 | 0 | 3
  Sarcoma | 1 | 1 | 0 | 0 | 2
  N/A | 0 | 0 | 17 | 14 | 31
  Missing | 3 | 4 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety--patients
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to measure anxiety in patient-participants. This scale is frequently used to assess psychosocial outcomes in cancer patients. The HADS is a 14-item self-report measurement tool designed for use in medical outpatient settings to assess depression and anxiety. Each subscale is scored from 0 to 21, with higher scores indicating greater distress; 0-7 is generally considered "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe" symptoms.
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in patients assigned to the intervention arm vs. patients assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS
Number analyzed (Participants) | 39 | 30
score on a scale | -1.4 (3.5) | -1.5 (2.7)
Statistical Analysis 1: Comparison: Intervention Arm--PATIENTS vs Wait List Control Arm--PATIENTS; Test type: Superiority; p = 1.00, ANOVA; Repeated measures ANOVA; F statistic = 0

2. Primary Outcome: Change in Depression--patients
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to measure depression in patients. This scale is frequently used to assess psychosocial outcomes in cancer patients. The HADS is a 14-item self-report measurement tool designed for use in medical outpatient settings to assess depression and anxiety. Each subscale is scored from 0 to 21, with higher scores indicating greater distress; 0-7 is generally considered "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe" symptoms.
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in patients assigned to the intervention arm vs. patients assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS
Number analyzed (Participants) | 39 | 31
score on a scale | -1.2 (3.1) | 0 (2.5)
Statistical Analysis 1: Comparison: Intervention Arm--PATIENTS vs Wait List Control Arm--PATIENTS; Test type: Superiority; p = 0.11, ANOVA; Repeated measures ANOVA; F statistic = 2.58

3. Primary Outcome: Change in Anxiety--caregivers
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to measure anxiety in caregiver-participants. This scale is frequently used to assess psychosocial outcomes in cancer patients. The HADS is a 14-item self-report measurement tool designed for use in medical outpatient settings to assess depression and anxiety. Each subscale is scored from 0 to 21, with higher scores indicating greater distress; 0-7 is generally considered "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe" symptoms.
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in caregivers assigned to the intervention arm vs. caregivers assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Number analyzed (Participants) | 12 | 12
score on a scale | -0.4 (3.2) | 0.3 (2.4)
Statistical Analysis 1: Comparison: Intervention Arm--CAREGIVERS vs Wait List Control Arm--CAREGIVERS; Test type: Superiority; p = 0.79, ANOVA; Repeated measures ANOVA; F statistic = 0.07

4. Primary Outcome: Change in Depression--caregivers
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to measure depression in caregiver-participants. This scale is frequently used to assess psychosocial outcomes in cancer patients. The HADS is a 14-item self-report measurement tool designed for use in medical outpatient settings to assess depression and anxiety. Each subscale is scored from 0 to 21, with higher scores indicating greater distress; 0-7 is generally considered "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe" symptoms.
Time Frame: Baseline to 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Number analyzed (Participants) | 12 | 12
score on a scale | -1.2 (2.0) | -0.3 (2.0)
Statistical Analysis 1: Comparison: Intervention Arm--CAREGIVERS vs Wait List Control Arm--CAREGIVERS; Test type: Superiority; p = 0.29, ANOVA; Repeated measures ANOVA; F statistic = 1.17

5. Secondary Outcome: Change in Distress--patients
Description: The National Comprehensive Cancer Network Distress Thermometer will be used to assess current distress level in patient-participants. Respondents are asked to rate their level of distress during the past week by circling a number on an image of a thermometer, with 0 indicating "no distress" and 10 "extreme distress".
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in patients assigned to the intervention arm vs. patients assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS
Number analyzed (Participants) | 40 | 31
score on a scale | -0.8 (3.2) | -0.5 (1.8)
Statistical Analysis 1: Comparison: Intervention Arm--PATIENTS vs Wait List Control Arm--PATIENTS; Test type: Superiority; p = 0.67, ANOVA; Repeated measures ANOVA; F statistic = 0.18

6. Secondary Outcome: Change in Fatigue--patients
Description: The Brief Fatigue Inventory assesses the severity and impact of cancer-related fatigue, asks about current level of fatigue, average and worst level of fatigue in the past 24 hours, and extent to which fatigue interfered with various aspects of life in the past 24 hours (e.g., mood, walking ability) on a 10-point Likert scale. A global fatigue score is calculated by averaging all items (ranging from 0 to 10). A higher score represents greater severity and impact of fatigue.
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in patients assigned to the intervention arm vs. patients assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS
Number analyzed (Participants) | 40 | 32
score on a scale | -0.8 (2.0) | 0 (1.5)
Statistical Analysis 1: Comparison: Intervention Arm--PATIENTS vs Wait List Control Arm--PATIENTS; Test type: Superiority; p = 0.24, ANOVA; Repeated measures ANOVA; F statistic = 1.41

7. Secondary Outcome: Change in Pain Interference--patients
Description: The 8-item Patient-Reported Outcomes Measurement Information System(PROMIS) pain interference scale will be used to measure the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Scores range from 8 to 40 with higher scores indicating more interference due to pain.
Time Frame: Baseline to 8 weeks
Population: Comparison of outcome in patients assigned to the intervention arm vs. patients assigned to the wait list control arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS
Number analyzed (Participants) | 30 | 20
score on a scale | -2.2 (8.3) | 0.8 (8.5)
Statistical Analysis 1: Comparison: Intervention Arm--PATIENTS vs Wait List Control Arm--PATIENTS; Test type: Superiority; p = 0.25, ANOVA; Repeated measures ANOVA; F statistic = 1.36

8. Secondary Outcome: Change in Distress--caregivers
Description: The National Comprehensive Cancer Network Distress Thermometer will be used to assess current distress level in caregiver-participants. Respondents are asked to rate their level of distress during the past week by circling a number on an image of a thermometer, with 0 indicating "no distress" and 10 "extreme distress".
Time Frame: Baseline to 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Number analyzed (Participants) | 13 | 12
score on a scale | -0.7 (2.2) | -0.2 (1.9)
Statistical Analysis 1: Comparison: Intervention Arm--CAREGIVERS vs Wait List Control Arm--CAREGIVERS; Test type: Superiority; p = 0.47, ANOVA; Repeated measures ANOVA; F statistic = 0.53

9. Secondary Outcome: Change in Fatigue--caregivers
Description: as for outcome 6
Time Frame: Baseline to 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Number analyzed (Participants) | 13 | 12
score on a scale | -0.8 (1.2) | -0.1 (1.6)
Statistical Analysis 1: Comparison: Intervention Arm--CAREGIVERS vs Wait List Control Arm--CAREGIVERS; Test type: Superiority; p = 0.23, ANOVA; Repeated measures ANOVA; F statistic = 1.54

10. Secondary Outcome: Change in Pain Interference--caregivers
Description: as for outcome 7
Time Frame: Baseline to 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
Number analyzed (Participants) | 9 | 8
score on a scale | 2.2 (4.6) | -0.4 (6.0)
Statistical Analysis 1: Comparison: Intervention Arm--CAREGIVERS vs Wait List Control Arm--CAREGIVERS; Test type: Superiority; p = 0.39, ANOVA; Repeated measures ANOVA; F statistic = 0.8

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Intervention Arm--PATIENTS: Patient participants in the intervention arm will receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks.
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Wait List Control Arm--PATIENTS: Patient participants in the wait list control arm will also receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks, but they will not receive access to the program until after the intervention group completes the intervention (8 weeks later).
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Intervention Arm--CAREGIVERS: Caregiver participants in the intervention arm will receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks.
  Mindfulness meditation program (administered via mobile app): Mobile app-based/online mindfulness meditation program
- Wait List Control Arm--CAREGIVERS: Caregiver participants in the wait list control arm will also receive access to a mobile app-based/online mindfulness meditation program and asked to practice meditation daily for 8 weeks, but they will not receive access to the program until after the intervention group completes the intervention (8 weeks later).
Arm/Group | Intervention Arm--PATIENTS | Wait List Control Arm--PATIENTS | Intervention Arm--CAREGIVERS | Wait List Control Arm--CAREGIVERS
All-Cause Mortality (participants affected / at risk) | 1/54 | 2/43 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/43 | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/54 | 0/43 | 0/17 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT03078608/Prot_SAP_000.pdf